CLINICAL TRIAL: NCT04862780
Title: A Phase 1/2 Study Targeting Acquired Resistance Mechanisms in Patients With EGFR Mutant Non-Small Cell Lung Cancer
Brief Title: (SYMPHONY) Phase 1/2 Study Targeting EGFR Resistance Mechanisms in NSCLC
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision, not related to safety concerns
Sponsor: Blueprint Medicines Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BLU-945-1101
Record Dates: First submitted 2021-04-21; First posted 2021-04-28 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Respiratory Tract Neoplasms; Neoplasms; Neoplasms by Site; Lung Diseases; Respiratory Tract Disease; Carcinoma, Bronchogenic; Bronchial Neoplasms; Adenocarcinoma; Carcinoma; Neoplasms by Histologic Type; Neoplasms, Nerve Tissue; EGFR T790M; EGFR C797S; EGFR L858R; EGFR Gene Mutation; EGF-R Positive Non-Small Cell Lung Cancer; EGFR Exon 19 Deletion; EGFR Mutation Resulting in Tyrosine Kinase Inhibitor Resistance; EGFR Activating Mutation; Protein Kinase Inhibitors; Antineoplastic Agents; Thoracic Neoplasms
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Respiratory Tract Neoplasms; Neoplasms; Neoplasms by Site; Lung Diseases; Respiratory Tract Diseases; Carcinoma, Bronchogenic; Bronchial Neoplasms; Adenocarcinoma; Carcinoma; Neoplasms by Histologic Type; Neoplasms, Nerve Tissue; Thoracic Neoplasms | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part 1A: BLU-945 as monotherapy (Experimental): Phase 1 dose escalation of BLU-945 as monotherapy at various dose levels
  Interventions: Drug: BLU-945
- Part 1B: BLU-945 with osimertinib (Experimental): Phase 1 dose escalation of BLU-945 in combination with osimertinib 80 mg tablets for oral administration
  Interventions: Drug: BLU-945; Drug: osimertinib
- Phase 2, Group 1: BLU-945 as monotherapy (Experimental): Phase 2 expansion group for BLU-945 as monotherapy at a dose determined during Part 1A in patients with EGFR T790M and C797S mutations
  Interventions: Drug: BLU-945
- Phase 2, Group 2: BLU-945 as monotherapy (Experimental): Phase 2 expansion group for BLU-945 as monotherapy at a dose determined during Part 1A in patients with EGFR T790M mutations
  Interventions: Drug: BLU-945
- Phase 2, Group 3: BLU-945 as monotherapy (Experimental): Phase 2 expansion group for BLU-945 as monotherapy at a dose determined during Part 1A in patients with EGFR C797S mutations
  Interventions: Drug: BLU-945
- Phase 2, Group 4: BLU-945 with osimertinib (Experimental): Phase 2 expansion group for BLU-945 with osimertinib at a dose determined during Part 1B in patients
  Interventions: Drug: BLU-945; Drug: osimertinib

INTERVENTIONS:
Drug: BLU-945 — Oral administration
Drug: osimertinib — Osimertinib tablets for oral administration
  Other Names: Tagrisso
  Arms: Part 1B: BLU-945 with osimertinib; Phase 2, Group 4: BLU-945 with osimertinib

SUMMARY:
This is a Phase 1/2, open-label, first-in-human (FIH) study designed to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and anticancer activity of BLU-945, a selective EGFR inhibitor, as monotherapy or in combination with osimertinib.

DETAILED DESCRIPTION:
The study will include an initial Phase 1 portion to determine the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of BLU-945 as monotherapy (initially in a QD regimen with the option to evaluate BID dosing, if supported by emerging PK and safety data), as well as an additional dose-escalation portion to determine the RP2D of BLU-945 in combination with osimertinib. The BLU-945 monotherapy Phase 2 expansion groups will consist of patients with tumors harboring specific mutation profiles (EGFR T790M and C797S mutation [Group 1]; EGFR T790M but not C797S [Group 2]; or EGFR C797S but not T790M [Group 3]). The BLU-945 with osimertinib Phase 2 expansion (Group 4) will include approximately 24 evaluable patients, with at least 12 slots reserved for patients with EGFR T790M and C797S mutation.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age at the time of signing the informed consent.
2. Pathologically confirmed, definitively diagnosed, metastatic NSCLC harboring an activating EGFR mutation.
3. Previously received at least 1 prior EGFR-targeted TKI with activity against the T790M mutation, such as osimertinib.

   a. Phase 1 Part 1B and Phase 2 Group 4: Patients must have experienced progressive disease while on osimertinib, and were able to tolerate prior osimertinib 80 mg QD dose.
4. Tumor mutation profile determined locally via a Sponsor-approved testing methodology, using tumor tissue (ideally from a progressing lesion) and/or ctDNA in plasma. For Phase 1, it is preferable that samples used for analysis be obtained during or after disease progression on the last EGFR-targeted TKI received. For Phase 2, pre-treatment tumor sample must be obtained during or after disease progression on the last EGFR-targeted TKI received.

   1. Dose Escalation (Phase 1 Part 1A and Part 1B): At each dose level, slots may be reserved for patients with the mutations of interest.
   2. BLU-945 Monotherapy Expansion Groups (Phase 2 Group 1, Group 2, and Group 3): Patients must have NSCLC harboring EGFR T790M and C797S mutation (Group 1); EGFR T790M but not C797S (Group 2); or EGFR C797S but not T790M (Group 3).
   3. BLU-945 with Osimertinib Expansion (Phase 2 Group 4): Slots may be reserved for patients with mutations of interest, but at least 12 slots will be allocated to patients with NSCLC harboring EGFR T790M and C797S mutation.
5. Pretreatment tumor sample (either an archival sample or a sample obtained by pretreatment biopsy) submitted for central analysis. For Phase 1, it is preferable that pretreatment tumor samples be obtained from a progression lesion, during or after disease progression on the last EGFR-targeted TKI received. For Phase 2, pre-treatment tumor sample must be obtained during or after disease progression on the last EGFR-targeted TKI received.

   Patients without appropriate archival tissue available, where biopsy is not considered safe and/or medically feasible, may be discussed with the study medical monitor and may be approved for enrollment on a case-by-case basis.
6. Phase 2 Expansion Groups: Patient has at least 1 measurable target lesion evaluable by RECIST 1.1 as assessed by the investigator.
7. Eastern Cooperative Oncology Group (ECOG) performance status is 0-1.
8. Agrees to use contraception consistent with the protocol and local regulations

Exclusion Criteria:

1. Tumor harbors any additional known driver alterations (including but not limited to EGFR exon 20 insertion, or pathologic abnormalities of KRAS, BRAF V600E, NTRK1/2/3, HER2, ALK, ROS1, MET, or RET).
2. NSCLC with mixed cell histology or a tumor with histologic transformation (NSCLC to SCLC, SCLC to NSCLC, or epithelial to mesenchymal transition).
3. Received the following anticancer therapy:

   1. EGFR-targeted TKI within 7 days prior to the first dose of study drug.
   2. Any immunotherapy or other antibody therapy (including EGFR-targeted antibodies or bi-specific antibodies) within 28 days prior to the first dose of study drug (immune-related toxicities must have resolved to < Grade 2 prior to starting BLU 945).
   3. Any other systemic anticancer therapy within 14 days or 5 half-lives prior to the first dose of study drug, whichever is the shortest, but with a minimum of 7 days in all circumstances. BLU 945 may be started within these washout periods if considered by the Investigator to be safe and within the best interest of the patient, with prior Sponsor approval.
   4. Radiotherapy to a large field or including a vital organ (including whole brain radiotherapy or stereotactic radiosurgery to brain) within 14 days before the first dose of study drug. Participant received radiotherapy to a focal site of disease that did not include a vital organ (such as a limb) within 7 days before the first dose of study drug.
4. CNS metastases or spinal cord compression that is associated with progressive neurological symptoms or requires increasing doses of corticosteroids to control the CNS disease. If a patient requires corticosteroids for management of CNS disease, the dose must have been stable for the 2 weeks preceding treatment. Asymptomatic CNS and leptomeningeal disease is allowed and, when measurable, should be captured as target lesions.
5. Any of the following abnormalities on the most recent laboratory test prior to the first dose of study drug (ie, Cycle 1 Day 1 [C1D1] or screening):

   1. Absolute neutrophil count (ANC) <1.0×109/L.
   2. Platelet count <75×109/L.
   3. Hemoglobin ≤8.0 g/dL (red blood cell transfusion and erythropoietin may be used to reach at least 8.0 g/dL, but must have been administered at least 2 weeks prior to the first dose of study drug).
   4. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >3× the upper limit of normal (ULN) if no hepatic metastases are present; >5× ULN if hepatic metastases are present.
   5. Total bilirubin >1.5× ULN; >3× ULN in presence of Gilbert's disease.
   6. Estimated (Cockroft-Gault formula) or measured creatinine clearance <40 mL/min.
   7. International normalized ratio (INR) >2.3 or prothrombin time (PT) >6 seconds above control or a patient-specific INR or PT abnormality that the treating investigator considers clinically relevant and/or increases the risk for hemorrhage in that individual patient.
6. Known intracranial hemorrhage and/or bleeding diatheses.
7. Clinically active ongoing interstitial lung disease (ILD) of any etiology, including drug-induced ILD, and radiation pneumonitis within 28 days prior to initiation of study treatment. Patients with prior ILD associated with clinically resolved COVID 19 infection may be enrolled upon discussion with, and approval by, the Medical Monitor.
8. Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 or that have not resolved to baseline at the time of starting the study. Exceptions include alopecia and fatigue, and, upon discussion with and approval by the Medical Monitor, other toxicities that are not thought to present a risk to patient safety.
9. Mean resting QT interval corrected using Fridericia's formula (QTcF) >450 msec, a history of prolonged QT syndrome or Torsades de pointes, or a familial history of prolonged QT syndrome.
10. Clinically significant, uncontrolled, cardiovascular disease including congestive heart failure Grade III or IV according to the New York Heart Association classification; myocardial infarction or unstable angina within the previous 6 months, uncontrolled hypertension, or clinically significant, uncontrolled arrhythmias, including bradyarrhythmia that may cause QT prolongation (eg, Type II second degree heart block or third-degree heart block).
11. History of another primary malignancy (other than completely resected carcinomas in situ) that has been diagnosed or required therapy within 2 years prior to initiation of study treatment. However, upon discussion with the Sponsor, the following categories of patients with prior malignancy are eligible to participate:

    1. Patients with a previous malignancy that completed all anticancer treatment at least 2 years before and with no evidence of residual disease from the prior malignancy at registration
    2. Patients who have another concurrent malignancy (not lung cancer) that is clinically stable and does not require tumor-directed treatment. (Examples include, but are not limited to, completely resected basal cell carcinoma and squamous cell carcinoma of skin, curatively treated prostate cancer, breast cancer and early gastric cancer cured by endoscopic mucosal resection or endoscopic submucosal dissection.)
12. Active, uncontrolled infection (viral, bacterial, or fungal) or active tuberculosis, hepatitis B, hepatitis C, AIDS-related illness, or known COVID 19 infection. Controlled infections, including HIV and "cured" hepatitis C (no active fever, no evidence of systemic inflammatory response syndrome) that are stable on antiviral treatment may be eligible if benefit/risk is justified and permission is granted from the Sponsor.
13. Dose-escalation (Parts 1A and 1B): Received neutrophil or platelet growth factor support within 14 days of the first dose of study drug.
14. Requires treatment with a prohibited medication or herbal remedy that cannot be discontinued at least 2 weeks before the start of study drug administration. BLU 945 may be started within 14 days or 5 half-lives of these therapies if considered by the Investigator to be safe and within the best interest of the patient, with prior Sponsor approval.
15. Major surgical procedure within 14 days of the first dose of study drug (procedures such as central venous catheter placement, tumor needle biopsy, and feeding tube placement are not considered major surgical procedures).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2024-10-07 (Actual); Study Completion 2024-10-07 (Actual)

PRIMARY OUTCOMES:
[Phase 1] Determine the maximum tolerated dose (MTD) of BLU-945 as monotherapy and BLU-945 in combination with osimertinib | Up to 12 months
  MTD determination: dose limiting toxicity (DLT) rate
[Phase 1] Rate and severity of adverse events of BLU-945 as monotherapy and BLU-945 in combination with osimertinib | Up to 12 months
[Phase 1] Determine recommended Phase 2 dose (RP2D) of BLU-945 as monotherapy and BLU-945 in combination with osimertinib | Up to 12 months
  RP2D determination: DLT, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary safety and anticancer activity data
[Phase 2] Overall response rate (ORR) of BLU-945 as monotherapy and BLU-945 in combination with osimertinib | Up to 30 months
  ORR, defined as the proportion of patients who experience a best response of confirmed CR or PR according to RECIST 1.1

SECONDARY OUTCOMES:
[Phase 1 and Phase 2] Cmax | Up to 42 months
[Phase 1 and Phase 2] Tmax | Up to 42 months
[Phase 1 and Phase 2] Tlast | Up to 42 months
[Phase 1 and Phase 2] AUC (0-24) | Up to 42 months
[Phase 1 and Phase 2] Ctrough | Up to 42 months
[Phase 1 and Phase 2] Vz/F | Up to 42 months
[Phase 1 and Phase 2] T 1/2 | Up to 42 months
[Phase 1 and Phase 2] CL/F | Up to 42 months
[Phase 1] Overall response rate (ORR) of BLU-945 as monotherapy and BLU-945 in combination with osimertinib | Up to 12 months
  ORR, defined as the proportion of patients who experience a best response of confirmed CR or PR according to RECIST 1.1
[Phase 1 and Phase 2] Duration of response (DOR) of BLU-945 as monotherapy and BLU-945 in combination with osimertinib | Up to 42 months
  DOR, defined as the time from first documented response of complete response (CR) or partial response (PR) to the date of first documented progressive disease or death due to any cause, whichever occurs first
[Phase 1 and Phase 2] Accumulation ratio | Up to 42 months
[Phase 1 and Phase 2] Assess treatment-induced modulation of EGFR pathway biomarkers. | Up to 42 months
  Profile pharmacodynamic changes in the EGFR pathway biomarker expression levels of dual specificity phosphatase (DUSP6) and sprouty RTK signaling antagonist 4 (SPRY4).
[Phase 2] Disease control rate (DCR) of BLU-945 as monotherapy and BLU-945 in combination with osimertinib | Up to 30 months
  DCR, defined as the proportion of patients who experience a best response of CR, PR, or stable disease (SD) according to RECIST 1.1
[Phase 2] Clinical benefit rate (CBR) of BLU-945 as monotherapy and BLU-945 in combination with osimertinib | Up to 30 months
  CBR, defined as the proportion of patients who experience a confirmed CR or PR, or stable disease (SD) with a duration of at least 16 weeks according to RECIST 1.1
[Phase 2] Progression free survival (PFS) of BLU-945 as monotherapy and BLU-945 in combination with osimertinib | Up to 42 months
  PFS, defined as the time from the first dose of BLU-945 until the date of first documented progressive disease or death due to any cause, whichever occurs first
[Phase 2] Overall survival (OS) of BLU-945 as monotherapy and BLU-945 in combination with osimertinib | Up to 42 months
  OS, defined as the time from the first dose of BLU-945 until the date of death due to any cause
[Phase 2] Central Nervous System Overall Response Rate (CNS-ORR) of BLU-945 as monotherapy and BLU-945 in combination with osimertinib | Up to 42 months
  CNS-ORR - proportion of patients with measurable (target) intracranial metastases at baseline who experience a confirmed intracranial CR or PR according to RECIST 1.1 principles
[Phase 2] Central Nervous System Duration of Response (CNS-DOR) of BLU-945 as monotherapy and BLU-945 in combination with osimertinib | Up to 42 months
  CNS-DOR - time from first documented intracranial CR or PR to the date of first documented intracranial PD
[Phase 2] Central Nervous System Progression Rate of BLU-945 as monotherapy and BLU-945 in combination with osimertinib | Up to 42 months
  CNS progression rate - proportion of patients with CNS progression as a component of first disease progression on study
[Phase 2] Rate and severity of adverse events of BLU-945 as monotherapy and BLU-945 in combination with osimertinib | Up to 42 months
[Phase 2] QTc Assessment | Up to 25 months
  Effects of BLU-945 on ECG parameters extracted from continuous 12 lead Holter recordings

CONTACTS AND LOCATIONS:
Locations (26):
- United States (10):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Cedars-Sinai Medical Center, Samuel Oschin Comprehensive Cancer Institute, Los Angeles, California
  - UC Irvine Health, Chao Family Comprehensive Cancer Center, Orange, California
  - University of Colorado Hospital - Anschutz Cancer Pavilion (ACP), Aurora, Colorado
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - NYU Langone Health, Laura and Isaac Perlmutter Cancer Center, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- France (2):
  - Institut Claudius Regaud (IUCT-O) - Cancer Comprehensive Center, Toulouse
  - Institut Gustave Roussy - DITEP, Villejuif
- Japan (3):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - National Cancer Center Hospital, Chuo Ku, Tokyo
- The Netherlands Cancer Institute - Antoni van Leeuwenhoek, Amsterdam, Netherlands
- National Cancer Centre Singapore, Singapore, Singapore
- South Korea (5):
  - Seoul National University, Department of Internal Medicine, Seoul
  - Yonsei Cancer Center, Severance Hospital, Yonsei University, Seoul
  - Asan Medical Center, Department of Oncology, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Vall d'Hebron University Hospital, Oncology Department, Barcelona, Spain
- National Taiwan University Hospital, Taipei, Taiwan
- The Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No